CLINICAL TRIAL: NCT04977154
Title: Prevention in Belgian Hockey : What Does the Staff Really Put in Place?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Gofflot Amandine, Principal Investigator, University of Liege
Other Study IDs: 160521
Record Dates: First submitted 2021-07-13; First posted 2021-07-26 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Primary Prevention; Questionnaire and Survey; Hockey Player
MeSH Terms: interventions — Primary Prevention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Trainers
  Interventions: Other: Primary prevention

INTERVENTIONS:
Other: Primary prevention — The primary prevention that the trainers put in place for the hockey players

SUMMARY:
Purpose: To provide an update on the implementation of prevention among hockey players by their entourage.

Materiel and method: This study will be conducted by the means of a questionnaire. The target population consisted of trainers.

The questionnaire will be validated by experts and published on an online survey website

ELIGIBILITY:
Inclusion Criteria:

* Professions: hockey trainer

Exclusion Criteria:

* /

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hockey trainer at different level of play
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Primary prevention by a questionnaire | Time Frame: The questionnaire will last 15 minutes at most
  The trainers will respond to a questionnaire that will inform us about the primary prevention that they put in place in hockey.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Liège, Liège, Belgium